CLINICAL TRIAL: NCT00433303
Title: Correlation Between Coital Activity During Pregnancy and Premature Delivery Related to Prostanoid Receptor Polymorphisms
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Other Study IDs: Intercourse-Prostanoid DP
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Last update posted 2007-02-09 (Estimated); Status verified 2007-02

CONDITIONS: Labor Onset; Gravidity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Correlation between early delivery and coital activity

SUMMARY:
The purpose of our study is correlate between premature delivery (between week 23-35 of the pregnancy) in women that had intercourse up to 12 hours prior to beginning of labor and polymorphisms in the gene Prostanoid receptor.

DETAILED DESCRIPTION:
During the past years there has been a conflict between different studies regarding the correlation between intercourse during pregnancy and early labor. Brustman et al showed that women that were at a high risk for early delivery and had intercourse and then an early labor had significantly increase uterine activity compared to women at low risk. Petridou et al showed that this risk is significantly higher at week 33 of gestation. However, the Cochrane Library summary leaves the question of correlation between intercourse and early labor unanswered. In Sayle et al's study showed no correlation between early delivery and intercourse. In 2004 Oguma described 3 polymorphisms in the Prostanoid receptor gene. These polymorphisms were correlated to increased activity of smooth muscles of bronchi in asthma. Since this gene is also expressed in the uterine muscles we wanted to determine whether there is a correlation between the three polymorphisms T-549C, C-441T, T-197C, G+1044A and early delivery due to intercourse.

1. Brustman LS, Raptoulis M. Langer O, Anyaegbunam A & Merkatz IR. Changes in the pattern of uterine contractility in relationship to coitus during pregnancies at low and high risk for preterm labor. Obstet Gynecol 1989;73:166-168
2. Petridou E, Salvnos H, Skalkidou A, Dessypris N, Moustaki M & Trichopoulos D. Are there common triggers of preterm deliveries. British J Obst Gynecol 2001;108:598-604)
3. Kavanagh J, Kelly AJ & Thomas J. Sexual intercourse for cervical ripening and induction of labour. The Cochrane Database of Systematic Reviews 2001, Issuse 2.Art. No.:CD003093. DOI: 10.1002/14651858.CD003093
4. Sayle AE, Savitz DA, Thorp JM, Hertz-Picciotto I & Wilcox AJ. Sexual activity during late pregnancy and risk of preterm delivery. Obstet Gynecol 2001;97:283-9)
5. Bernal AL. Mechanisms of labour-biochemical aspects. BJOG 2003;110(Supp 20):39-45
6. Oguma T, Palmer L, Birden E, Sonna LA, Asano K& Lilly CM. Role of prostanoid dp receptor variants in susceptibility to asthma. NEJM 2004;351:1752-63

ELIGIBILITY:
Inclusion Criteria:

* Women who start delivery in weeks 23-35 of pregnancy 12 hours after intercourese.
* Women who come for delivery after week 31 and have not had intercourse during the previous month.
* Women at term who have been sexually active during their pregnancy.

Exclusion Criteria:

* Any other women who come in for delivery.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schimmel, Prof., Principal Investigator — Neonatology Unit, Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Brustman LE, Raptoulis M, Langer O, Anyaegbunam A, Merkatz IR. Changes in the pattern of uterine contractility in relationship to coitus during pregnancies at low and high risk for preterm labor. Obstet Gynecol. 1989 Feb;73(2):166-8. PMID 2911421